CLINICAL TRIAL: NCT00991445
Title: Minimal vs. Conventional Exposure in Unicompartmental Knee Arthroplasty
Brief Title: Minimal Versus Conventional Exposure in Unicompartmental Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Professor Kjell Axelsson, University Hospital Orebro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAK-Incision
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Knee Osteoarthritis
Keywords: Unicompartmental knee arthroplasty; Surgical exposure; Minimal invasive surgery; Local Infiltration Analgesia; Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group MIS (Active Comparator): Minimal Invasive Surgery
  Interventions: Procedure: Minimal Invasive Surgery
- Conventional Exposure (Active Comparator)
  Interventions: Procedure: Conventional exposure

INTERVENTIONS:
Procedure: Minimal Invasive Surgery — After a 8-10 cm skin incision, a medial parapatellar capsule incision is made. The vastus medialis muscle or the rectus tendon are not incised, nor is the patella everted. The patella is merely pushed slightly aside when the bone cuts are made and the prostheses are cemented in place. Local Infiltration Analgesia is used.
  Arms: Group MIS
Procedure: Conventional exposure — After a 15-20 cm midline skin incision is made, a medial parapatellar capsule incision is made. The incision is carried up through the insertion of the vastus medialis and into the rectus tendon. The patella is everted. The bone cuts are made and the prostheses are cemented in place. Local Infiltration Analgesia is used.
  Arms: Conventional Exposure

SUMMARY:
The purpose of this study is to determine whether Minimal Invasive Surgery results in less postoperative pain and better mobilization than conventional technique in Unicompartmental Knee Arthroplasty, provided that both groups receive Local Infiltration Analgesia.

DETAILED DESCRIPTION:
Postoperative pain is often moderate to severe following unicompartmental knee arthroplasty. In order to reduce postoperative pain and improve mobilization the minimal invasive technique was developed. After a 8-10 cm skin incision, a medial parapatellar capsule incision in made. The rectus tendon or the vastus medialis are not incised and the patella is not everted.

In recent years The Local Infiltration Analgesia (LIA) technique has been developed to reduce postoperative pain. With this LIA-technique, a long-acting local anesthetic (ropivacaine), a nonsteroidal anti-inflammatory drug (ketorolac), and epinephrine are infiltrated intraoperatively and via an intraarticular catheter postoperatively.

The aim of this study is to investigate if Minimal Invasive Surgery results in less postoperative pain and better mobilization than conventional technique in Unicompartmental Knee Arthroplasty, provided that both groups receive Local Infiltration Analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for unicompartmental knee arthroplasty
* Aged 20-80 yrs
* ASA physical status I-III and mobility indicating normal postoperative mobilization

Exclusion Criteria:

* Known allergy or intolerance to local anesthetics, ASA or NSAID
* Serious liver-, heart- or renal decease
* Rheumatoid arthritis
* Chronic pain or bleeding disorder

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Time to fulfilling discharge criteria | 0-2 weeks

SECONDARY OUTCOMES:
Pain intensity | 0-3 months
Hospital stay | 0-2 weeks
Morphine consumption | 0-48 hours
Knee function | 0-3 months
Patient satisfaction | 0-3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Axelsson, Professor, Principal Investigator — Region Örebro County
Locations (1):
- Dept. of Orthopedic Surgery, Örebro, Örebro County, Sweden

REFERENCES:
- [Derived] Essving P, Axelsson K, Otterborg L, Spannar H, Gupta A, Magnuson A, Lundin A. Minimally invasive surgery did not improve outcome compared to conventional surgery following unicompartmental knee arthroplasty using local infiltration analgesia: a randomized controlled trial with 40 patients. Acta Orthop. 2012 Dec;83(6):634-41. doi: 10.3109/17453674.2012.736169. Epub 2012 Oct 8. PMID 23043272